CLINICAL TRIAL: NCT01393938
Title: Comparison of MRI Versus Three Dimensional Ultrasound in the Diagnosis of Mullerian Duct Anomalies
Acronym: MDA-3DUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN090691BE2010
Record Dates: First submitted 2011-05-27; First posted 2011-07-13 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Mullerian Duct Anomaly
Keywords: Mullerian Duct Anomaly; 3-dimensional Ultrasound; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mullerian Duct Anomaly (Other)
  Interventions: Other: Three-dimensional ultrasound

INTERVENTIONS:
Other: Three-dimensional ultrasound — Immediately following the standard of care 2D-US, for approximately 15 min.

SUMMARY:
Mullerian duct anomalies (MDAs) are relatively common disorders, with a prevalence estimated to be around 2% in the general population, and 6% to 7% in women with a history of recurrent pregnancy loss. Mullerian duct anomalies are associated with recurrent pregnancy loss, intra uterine growth retardation, and preterm labor and birth. The prevalence of preterm birth and pregnancy loss varies with the type of MDA. Patients can benefit from surgery or hysteroscopic interventions like metroplasty based on the type of MDA. Therefore, to optimize patient outcomes, accurate diagnosis and description of MDAs is essential.

Magnetic resonance imaging (MRI) is an excellent way of evaluating the uterus for MDAs. MRI, although costly, is less expensive than laparoscopy and hysteroscopy and is non-invasive. Pellerito et all evaluated 26 women with surgically proven MDAs and found that in 24 cases MRI was able to correctly diagnose the MDAs. Therefore MRI is generally considered as a reference standard for uterine evaluation. In a study comparing MRI and endovaginal Two-Dimensional Ultrasound (2DUS), MRI appeared to be more accurate than 2DUS with a sensitivity of 77%, specificity of 33%, and a positive predictive value of 83%.

Endovaginal Three-Dimensional Ultrasound (3DUS) is a relatively new technology that creates three-dimensional volumes from a series of two-dimensional images. This technique allows the user to acquire coronal or face-on-view of the uterus which is essential in evaluating the uterus for the presence of MDAs. Kupesic and Kurjak used 3DUS to evaluate 86 patients and found that it had sensitivity of 98.38%, specificity of 100%, a positive predictive value of 100%, and a negative predictive value of 96% in the diagnosis of septate uteri [7]. Endovaginal 3DUS is less expensive, less invasive, and less-time consuming than hysteroscopy or MRI and appears to be a very promising technology for the evaluation of MDAs. 3DUS appears to be at least as accurate as MRI in the diagnosis of MDAs. In addition, 3DUS is less expensive than MRI and in some patients better tolerated. If validated using prospective studies, 3DUS has the potential to become the reference standard for the diagnosis of MDAs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16
2. Patients with suspected Mullerian Duct Anomalies (history of recurrent miscarriage or history of primary or secondary infertility).
3. Patients scheduled to undergo routine endovaginal or transabdominal Ultrasonography and pelvic MRI to evaluate possible MDAs

Exclusion Criteria:

1. Age < 16
2. General contraindications to MRI such as pacemaker etc.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of 3D US and MRI in the diagnosis and assessment of patients with MDAs | US and MRI within 1 month
  Currently the best way for imaging Müllerian Duct Anomalies (MDAs) is Magnetic Resonance Imaging (MRI). In addition, doctors use Two Dimensional Ultrasound (2D-US) to obtain additional pictures of these abnormalities.
  Three Dimensional Ultrasound is a new imaging method recently being used to assess these abnormalities. It works in exactly the same way as 2D-US, the only difference being a more up to date computer software, which helps obtain the better images.
  This study will assess the accuracy of MRI versus Three Dimensional Ultrasound in viewing and correctly diagnosing MDAs.

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada